CLINICAL TRIAL: NCT01477151
Title: Randomized Isoflurane and Sevoflurane Comparison in Cardiac Surgery: A Prospective Randomized Clinical Trial.
Brief Title: Randomized Isoflurane and Sevoflurane Comparison in Cardiac Surgery
Acronym: RISCCS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Philip Jones, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16497
Record Dates: First submitted 2011-11-16; First posted 2011-11-22 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Coronary Artery Disease; Valvular Heart Disease
Keywords: isoflurane; sevoflurane; troponin; anesthesia; cardioprotection; preconditioning; cardiac surgery; cardiac anesthesia
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sevoflurane (Active Comparator): These patients will receive sevoflurane as the volatile anesthetic pre-, during-, and post-cardiopulmonary bypass at a targeted dose of 0.5-2.0 MAC.
  Interventions: Drug: Volatile anesthetic
- isoflurane (Experimental): These patients will receive isoflurane as the volatile anesthetic pre-, during-, and post-cardiopulmonary bypass at a targeted dose of 0.5-2.0 MAC.
  Interventions: Drug: Volatile anesthetic

INTERVENTIONS:
Drug: Volatile anesthetic — The intervention in this trial is randomization to either maintenance of anesthesia with sevoflurane or maintenance of anesthesia with isoflurane. The designated volatile anesthetic will be given at a strict minimal amount throughout the entire cardiac surgery (including cardiopulmonary bypass). This regimen (administration throughout the entire operation) has proved to have the greatest efficacy. Apart from this intervention, the anesthetic for patients participating in this trial will not be substantially different from normal practice, as the intention is to allow normal practice (with the exception of the choice of volatile anesthetic agent) to maximize the applicability and external validity of the trial. The management of anticoagulation, cardiac surgical techniques, and other aspects of the procedure will be managed in an unaltered fashion.
  No IV drug infusions will be permitted until after protamine administration.

SUMMARY:
Anesthesia practice in the 21st century is increasingly outcomes-oriented and evidence-based, but there remain significant gaps in our knowledge, even for commonly-encountered clinical situations. Currently, the two most commonly used drugs used for maintenance of anesthesia in cardiac surgical patients are isoflurane and sevoflurane. There is a belief among many cardiac anesthesiologists that sevoflurane is a better cardiac anesthetic than isoflurane, but there is very little data to support this notion. In fact, very little is known about their comparative effects on important patient outcomes because there has not been a large head-to-head prospective randomized clinical trial. This project will supply the data necessary to critically compare the two anesthetics.

DETAILED DESCRIPTION:
Current evidence supports the superiority of sevoflurane for myocardial protection during cardiac surgery when compared to total intravenous anesthesia with propofol. However, there is no evidence to suggest that sevoflurane is superior to isoflurane for myocardial protection during cardiac surgery. Sevoflurane may potentially reduce the rate of post-cardiac surgery atrial fibrillation and the time to tracheal extubation compared to isoflurane, but the literature is equivocal on these two important outcomes. Anesthesiologists still frequently use isoflurane for maintenance of cardiac anesthesia, and this is likely because there is substantial uncertainty about whether or not sevoflurane is superior to isoflurane, given the lack of head-to-head RCTs. A large, prospective, pragmatic RCT can ultimately assist clinicians by providing evidence of the non-inferiority (or, possibly the superiority) of one anesthetic compared to the other on important patient outcomes such as ICU length of stay, mortality, renal dysfunction, time to tracheal extubation after cardiac surgery, rates of clinically-important atrial fibrillation, and myocardial damage.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years or over (There is no upper age limit to enrollment)
* Eligible procedures are: CABG on-pump or off-pump, single valve repair/replacement, or CABG/single valve combined procedures

Exclusion Criteria:

* Cardiac surgeries that are not one of the included cases
* Planned extubation in the operating room
* Patients refusing blood products (vis à vis blood sampling)
* Pregnant patients
* Malignant hyperthermia or documented/stated allergy to potent volatile anesthetic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2011-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Composite of: prolonged ICU stay (>= 48 hours) OR death within 30 days of operation | 30 days of operation

SECONDARY OUTCOMES:
Postoperative cardiac troponin T | 6 hours after admission to ICU
  Troponin T sampled at 6 hours after admission to the ICU. The time of sampling will be recorded. The sample will be taken from an indwelling venous or arterial cannula (if one exists) or by venipuncture.
Length of stay in the ICU (criteria) | Participants will be followed for the duration of ICU stay, an expected average of 1 day
  The time from admission in ICU (time 0) until the patient's transfer orders to the floor are enacted.
30-day all-cause mortality | 30 days after operation
  A participant who has died for any reason before the end of 30th day after the operation. Day 1 is the first calendar day after first being admitted to the ICU.
Duration of tracheal intubation | Participants will be followed for the duration of ICU stay, an expected average of 1 day
  The time from being admitted to the ICU (time 0) until the patient's tracheal tube is removed for the first time.
Inotrope or vasopressor usage in the ICU | Participants will be followed for the duration of ICU stay, an expected average of 1 day
  A participant who is treated at any time after the first hour of their ICU stay with an inotropic or vasopressor by infusion.
Prolonged inotrope or vasopressor usage in the ICU | Participants will be followed for the duration of ICU stay, an expected average of 1 day
  Any patient requiring 12 or more continuous hours of any combination of inotropic or vasopressor agent (including the first hour) in the ICU.
Peak postoperative serum creatinine | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Peak postoperative creatinine as recorded in the hospital chart.
New-onset dialysis | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Any patient, not previously on dialysis, requiring postoperative dialysis (hemodialysis or peritoneal dialysis).
Incidence of new-onset atrial fibrillation | Until end of post-operative day 4
  We will capture the proportion of patients who have clinically significant new atrial fibrillation at any time from ICU admission until the end of POD 4. The adjudication of atrial fibrillation will be recorded by the blinded research nurse.
Incidence of intra-aortic balloon pump usage | Participants will be followed for the duration of ICU stay, an expected average of 1 day
  The proportion of patients having an intra-aortic balloon pump inserted (either in the operating room or in the ICU).
Length of stay in the ICU (actual) | Participants will be followed for the duration of ICU stay, an expected average of 1 day
  The time from admission in ICU (time 0) until the patient is discharged from the ICU.
Length of stay in the hospital (actual) | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  The time from admission to the ICU until the patient is discharged home from the hospital.
Readmission to ICU | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Readmission to the ICU for any reason.
Perioperative stroke | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  A new neurological abnormality persisting > 24 hours with documentation by formal neurological examination and evidence of new brain lesions on a brain imaging study.
1-year all-cause mortality | One year after operation
  A participant who has died for any reason within the first year after the operation. For example, if the operation takes place on June 20 2011, then mortality up to and including June 19 2012 will be counted.

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Jones, MD MSc, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- University Hospital - London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Jones PM, Bainbridge D, Chu MWA, Fernandes PS, Fox SA, Iglesias I, Kiaii B, Lavi R, Murkin JM. Comparison of isoflurane and sevoflurane in cardiac surgery: a randomized non-inferiority comparative effectiveness trial. Can J Anaesth. 2016 Oct;63(10):1128-1139. doi: 10.1007/s12630-016-0706-y. Epub 2016 Jul 27. PMID 27465213